CLINICAL TRIAL: NCT02824731
Title: Comparison of Proton and Photon Radiotherapy of Brain Tumors: Efficiency and Side Effects in Clinical Standard Doses
Brief Title: Comparison of Proton and Photon Radiotherapy of Brain Tumors (ProtoChoice-Hirn)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: German Cancer Research Center (Other); National Center for Radiation Research in Oncology Dresden/Heidelberg (Other)
Responsible Party: Principal Investigator, Mechthild Krause, Principal Investigator, Technische Universität Dresden
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STR - ProtoChoice-Hirn - 2015
Record Dates: First submitted 2016-05-11; First posted 2016-07-07 (Estimated); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Brain Tumors
Keywords: brain tumors; proton radiotherapy; photon radiotherapy
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiation; Protons; Photons

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- supratentorial, grade III/IV, photon (Active Comparator): Radiation with photons normofractionated 54-60 Gy. Not pre-irradiated patients.
  Interventions: Radiation: Radiation with photons
- supratentorial, grade III/IV, proton (Experimental): Radiation with protons normofractionated 54-60 Gy(RBE). Not pre-irradiated patients.
  Interventions: Radiation: Radiation with protons
- supratentorial, grade I/II, photon (Active Comparator): Radiation with photons normofractionated 54-60 Gy. Not pre-irradiated patients, bening tumors.
  Interventions: Radiation: Radiation with photons
- supratentorial, grade I/II, proton (Experimental): Radiation with protons normofractionated 54-60 Gy(RBE). Not pre-irradiated patients, bening tumors.
  Interventions: Radiation: Radiation with protons
- infratentorial, photon (Active Comparator): Radiation with photons normofractionated 54-60 Gy. Not pre-irradiated patients.
  Interventions: Radiation: Radiation with photons
- infratentorial, proton (Experimental): Radiation with protons normofractionated 54-60 Gy(RBE). Not pre-irradiated patients.
  Interventions: Radiation: Radiation with protons
- pre-radiation, photon (Active Comparator): > 40Gy in the region of recurrence. Radiation with photons normofractionated 54-60 Gy(RBE) or 5 Gy(RBE)/fraction until 30 Gy(RBE) or normofractionated 36 Gy(RBE).
  Interventions: Radiation: Radiation with photons
- pre-radiation, proton (Experimental): > 40Gy in the region of recurrence. Radiation with protons normofractionated 54-60 Gy(RBE) or 5 Gy(RBE)/fraction until 30 Gy(RBE) or normofractionated 36 Gy(RBE).
  Interventions: Radiation: Radiation with protons

INTERVENTIONS:
Radiation: Radiation with protons
  Arms: infratentorial, proton; pre-radiation, proton; supratentorial, grade I/II, proton; supratentorial, grade III/IV, proton
Radiation: Radiation with photons
  Arms: infratentorial, photon; pre-radiation, photon; supratentorial, grade I/II, photon; supratentorial, grade III/IV, photon

SUMMARY:
This protocol compares the toxicity of radiotherapy or radiochemotherapy applied with different radiation modalities - protons or photons. Patients with different kinds of brain tumours and foreseen high-dose radiotherapy can be included. The hypothesis of the trial is that the rate of chronic toxicity 1 year after the end of radiotherapy is 15% lower after proton compared to photon treatment.

DETAILED DESCRIPTION:
Non-randomised 2-arm phase II trial on comparison of proton versus photon radiotherapy in brain tumours using standard doses and standard combined chemotherapy protocols. Patients are assigned to the treatment groups by their own choice or availability of the treatment. Patients are stratified into 4 groups, (1) supratentorial grad III/ IV tumours without pre-irradiation; (2) supratentorial grade I/II tumours without pre-irradiation; (3) infratentorial tumours without pre-irradiation; (4) patients with pre-irradiation >40 Gy in the tumour area. Radiotherapy doses of 54-60 Gy(RBE) are applied in group 1-3 using normal fractionated schedules. In group 4, 30 Gy(RBE)/ 5 Gy(RBE) per fraction or 36 Gy(RBE) with 2 Gy(RBE) per fraction are allowed. Primary endpoint is chronic toxicity and quality of life. The hypothesis of the trial is that the rate of chronic toxicity 1 year after the end of radiotherapy is 15% lower after proton compared to photon treatment. Events for chronic toxicity are toxicities observed later than 3 months after end of radiotherapy and scored CTC-AE4.0 >grade 2 or a decrease in Quality of life by >10% (EORTC-QLQ C30 and BN20) or a decrease in neuropsychological functioning by >10% (MoCa test). All statistical calculations apply to group (1), i.e. supratentorial grade II/IV tumours without pre-irradiation, all other arms are closed when group (1) is closed.

ELIGIBILITY:
Inclusion Criteria:

* primary brain tumor: gliomas (low or high grade), intracerebral meningiomas, pituitary adenomas, craniopharyngioma and other rare brain tumors or
* brain tumor recurrence without pre-irradiation or
* brain tumor recurrence with pre-irradiation > 40 Gy in the overlap region with the recurrence region
* indication for radiotherapy or radiochemotherapy
* Both proton and photon therapy are possible from a medical point of view (that is no standard indication for protons or standard indication for example one-time stereotaxy
* age >= 18 years
* general condition ECOG ≤ 2, outpatient basis possible
* indication for high dose (except group 4) radiotherapy or radiochemotherapy
* capacity to consent and present written informed consent

Exclusion Criteria:

* lack of capacity to consent or lack of written consent
* cerebral lymphomas
* brain metastases
* very small tumors (for example acoustic neuromas, very small recurrences) for this is a proton therapy from a medical point of view no alternative to a stereotactic radiotherapy
* inability to MRI planning (eg. contraindications to performing MRI)
* lack of compliance of the patient
* lack of or limited possibility of a reproducible storage (eg by severe restriction of mobility of the patient)
* missing or limited possibility of regular follow-up visits in accordance with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 555 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
late toxicity as cumulative measure | 1 year (or at least 6 months)
  Events for the endpoint are:
  1. any late toxicity CTCAE 4.0 ≥ grade II (except pre-existing conditions)
  2. decrease in Quality of life (EORTC-QLQ-C30 and BN20) by >10%
  3. decrease in brain function (MOCA test) by more than 10%

SECONDARY OUTCOMES:
Local tumour control | 1 year and 2 years
  Local tumour control as Regression or stable disease measured in follow-up MRI
Overall survival | 1 year and 2 years
  Overall survival
Acute toxicity | 3 months after treatment
  Acute toxicity according to CTCAE4.0 score >/= grade II
late toxicity as cumulative measure | 2 years
  Events for the endpoint are:
  1. any late toxicity CTCAE 4.0 ≥ grade II (except pre-existing conditions)
  2. decrease in Quality of life (EORTC-QLQ-C30 and BN20) by >10%
  3. decrease in brain function (MOCA test) by more than 10%

CONTACTS AND LOCATIONS:
Overall Officials: Mechthild Krause, Prof., Study Chair — University of Technology, University Hospital Carl Gustav Carus, Department of Radiation Therapy and Radiation Oncology, German Consortium for Translational Cancer Research (DKTK)
Locations (2):
- Germany (2):
  - University Hospital Carl Gustav Carus, Department of Radiotherapy and Radiation Oncology, Dresden
  - University Hospital Gießen and Marburg, Department of Radiotherapy and Radiation Oncology, Marburg

IPD SHARING:
Plan to Share IPD: No